CLINICAL TRIAL: NCT01367223
Title: Modulation of Systemic Inflammatory Response in Critically Ill Children After Glutamine Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Sant Joan de Deu (Other)
Collaborators: Fundació Sant Joan de Déu (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCIHSJD5
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Inflammatory Response; Multi-organ Failure
Keywords: inflammatory response; parenteral nutrition; glutamine; amino acid; pediatric; intensive care; systemic infection; abdominal surgery; polytraumatised; mortality; mean stay in the intensive care unit; occurrence of infections
MeSH Terms: conditions — Multiple Organ Failure; Hyperphagia; Toxemia | interventions — Glutamine; amino-acid, glucose, and electrolyte solution; alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- solution of amino acids with glutamine (Experimental): Group 1 as the experimental group who will be administered a solution of amino acids supplemented with glutamine
  Interventions: Dietary Supplement: solution of amino acids supplemented with glutamine
- amino acids solution without glutamine (Other): Group 2:control group will be administered a solution of amino acids (Aminoven Infant® or Vamin®) not supplemented with glutamine
  Interventions: Dietary Supplement: amino acids not supplemented with glutamine

INTERVENTIONS:
Dietary Supplement: solution of amino acids supplemented with glutamine — parenteral nutrition by range of ages (recommendation from ESPGHAN and ESPEN:1 month to 3 years, 3 to 5 years, 6 to 12 and standard adult).Study Parenteral nutrition will be assessed the first 5 days.
  Other Names: (Aminoven Infant® or Vamin®) with glutamine (Dipeptiven®)
  Arms: solution of amino acids with glutamine
Dietary Supplement: amino acids not supplemented with glutamine — parenteral nutrition by range of ages (recommendation from ESPGHAN and ESPEN:1 month to 3 years, 3 to 5 years, 6 to 12 and standard adult).Study Parenteral nutrition will be assessed the first 5 days.
  Other Names: (Aminoven Infant® or Vamin®) with glutamine (Dipeptiven®)
  Arms: amino acids solution without glutamine

SUMMARY:
This study aims to describe the use of glutamine supplementation in the modulation of inflammatory response in critically ill pediatric patients and to determine if this decrease leads to clinical improvement in morbidity and mortality in these patients. Thus, these patients' diet could be supplemented with glutamine in order to improve their evolution.

Hypothesis:

From the data obtained in the study of the literature the investigators consider that:

Critically ill patients have a deficit of glutamine either because of an increase in its consumption or a decrease in its availability, and therefore blood glutamine levels are low.

Critically ill patients have elevated blood levels of pro-inflammatory substances (IL-6).

In these patients tissue lesion inhibitors (HSP-70) in the blood are decreased. The administration of glutamine supplements to these patients decreases oxidative stress due to the increase in HSP-70.

Inflammation inhibitory substances (IL-10) in the blood are decreased in these patients.

The administration of glutamine supplements in these patients increase IL-10 levels.

Glutamine supplements decrease the inflammatory response with a decrease in IL-6 levels.

DETAILED DESCRIPTION:
Objective

This study aims to describe the use of glutamine supplementation in the modulation of inflammatory response in critically ill pediatric patients and to determine if this decrease leads to clinical improvement in morbidity and mortality in these patients. Thus, these patients' diet could be supplemented with glutamine in order to improve their evolution.

In recent years numerous studies have been conducted and published on the different factors, amongst them glutamine, that could modulate the inflammatory response of critically ill patients thus reducing the impact this response has and its progression to multi-organ failure.

Glutamine (Gln) is the most abundant amino acid in the body and is mainly synthesised in skeletal muscle. It is a non-essential amino acid that is produced is sufficient quantities in good states of health. Plasma levels are above 0.6 mmol/L, and 50% is found in the free form in plasma1. This amino acid not only acts as a source of energy but it is also involved in the synthesis of other amino acids, nucleotides, nucleic acids, sugars, amines, proteins and different biologically active molecules2. Other functions are: maintenance of the internal acid-base homeostasis, urea synthesis, glyconeogenesis, neurotransmission, and cell differentiation and proliferation. It is also the main energy substrate for the rapidly proliferating cells (enterocytes) and of multiple immune cells (macrophages, monocytes, lymphocytes). It also takes part in the protection of cells and tissues inducing expression of the heat shock proteins3.

In recent years, numerous studies have been performed to determine the effect of Gln, both by enteral and parenteral route, on the evolution of critically ill patients. These studies were conducted in animals and in humans, mainly adults. However, there is little reference in the literature to studies in children. The studies are based on the use of glutamine as a dietary supplement mainly in patients with neoplastic disease or inflammatory bowel disease. It has also been studied as a supplement in premature infants, but there are very few studies in critically ill children.

In the last year many studies have been published on the use of glutamine. The effect of glutamine supplementation on the intestinal mucosal barrier in rabbits under haemorrhagic shock was studied. Shock was induced by blood withdrawing from the femoral artery; the rabbits were randomised to three groups (control, low dose glutamine and high dose glutamine). Plasma levels of diamine oxidase and IL-8 were measured and a histological examination of the terminal ileum was performed. The results demonstrated a lower inflammatory and oxidative response in the rabbits who had received Gln supplementation37. Another study in rats measured the effect of the dipeptide Arginin - Gln on endothelial cell growth factor levels in retinal pigment epithelial cell cultures and on the inhibition of neovascularisation in oxygen-induced retinopathy. The authors concluded that they decreased with the administration of this dipeptide38. Another factor studied in critically ill patients was the oxidative activity measured as diamine oxidase activity and D-lactate content39. Protection against infection and decrease in insulin resistance in critically ill patients is still being studied 21,22, 32, 40, 41. Contradictory findings have been reported therefore new studies are required in systematic reviews.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 1 month and 14 years who require parenteral nutrition according to the criteria of our unit and who comply with the following diagnoses:

* Local or systemic infection
* Post abdominal surgery
* Polytraumatised

Parenteral nutrition indications:

* Intestinal resections
* Bowel obstruction or post-surgery
* Risk of intestinal ischaemia due to hypotension of hypoxaemia

Exclusion Criteria:

1. Legal representative does not give consent.
2. Patients with previous underlying diseases (renal impairment, hepatic impairment, inflammatory bowel disease, rheumatic diseases, metabolic diseases, immunocompromised).
3. Mild liver impairment on admittance (hepatitis, colostasis).
4. Post cardiac surgery with extracorporeal circulation.
5. Patients referred from other hospitals with a clinical evolution of over 48 hours.
6. Patients aged less than one month and over 14 years.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint is to determine if there are any differences in inflammatory response in patients supplemented with glutamine compared to those who receive a standard diet without a glutamine supplement. | baseline-day2-day5
  Laboratory measures: IL-6, IL-10, HSP-70

SECONDARY OUTCOMES:
As secondary endpoints the clinical response of the two groups of patients was assessed with respect to the occurrence of infections, multi-organ failure, mean stay in the unit and mortality. | During 27 days

CONTACTS AND LOCATIONS:
Overall Officials: Iolanda Jordan, PhMD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Bracco D. Glutamine: a double edge sword in the intensive care unit? Crit Care Med. 2005 Nov;33(11):2692-4. doi: 10.1097/01.ccm.0000186750.06199.0f. No abstract available. PMID 16276205
- [Background] Yeh CL, Hsu CS, Yeh SL, Chen WJ. Dietary glutamine supplementation modulates Th1/Th2 cytokine and interleukin-6 expressions in septic mice. Cytokine. 2005 Sep 7;31(5):329-34. doi: 10.1016/j.cyto.2005.06.001. PMID 16026997
- [Background] Wischmeyer PE. Can glutamine turn off the motor that drives systemic inflammation? Crit Care Med. 2005 May;33(5):1175-8. doi: 10.1097/01.ccm.0000162686.28604.81. No abstract available. PMID 15891373
- [Background] Fuentes-Orozco C, Anaya-Prado R, Gonzalez-Ojeda A, Arenas-Marquez H, Cabrera-Pivaral C, Cervantes-Guevara G, Barrera-Zepeda LM. L-alanyl-L-glutamine-supplemented parenteral nutrition improves infectious morbidity in secondary peritonitis. Clin Nutr. 2004 Feb;23(1):13-21. doi: 10.1016/s0261-5614(03)00055-4. PMID 14757388
- [Background] Schulman AS, Willcutts KF, Claridge JA, O'Donnell KB, Radigan AE, Evans HL, McElearney ST, Hedrick TL, Lowson SM, Schirmer BD, Young JS, Sawyer RG. Does enteral glutamine supplementation decrease infectious morbidity? Surg Infect (Larchmt). 2006 Feb;7(1):29-35. doi: 10.1089/sur.2006.7.29. PMID 16509783
- [Background] Tubman TR, Thompson SW, McGuire W. Glutamine supplementation to prevent morbidity and mortality in preterm infants. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001457. doi: 10.1002/14651858.CD001457.pub2. PMID 15674878
- [Background] Coeffier M, Dechelotte P. The role of glutamine in intensive care unit patients: mechanisms of action and clinical outcome. Nutr Rev. 2005 Feb;63(2):65-9. doi: 10.1111/j.1753-4887.2005.tb00123.x. PMID 15762090
- [Background] Deutschman CS, Levy RJ, Weiss YG. Glutamine and heat shock proteins: one more approach to lung injury. Crit Care Med. 2005 Jun;33(6):1422-4. doi: 10.1097/01.ccm.0000167072.03551.61. No abstract available. PMID 15942367
- [Background] Choudhry MA, Haque F, Khan M, Fazal N, Al-Ghoul W, Ravindranath T, Gamelli RL, Sayeed MM. Enteral nutritional supplementation prevents mesenteric lymph node T-cell suppression in burn injury. Crit Care Med. 2003 Jun;31(6):1764-70. doi: 10.1097/01.CCM.0000063053.31485.DF. PMID 12794418
- [Background] Andrews F, Griffiths R. Glutamine-enhanced nutrition in the critically ill patient. Hosp Med. 2002 Mar;63(3):144-7. doi: 10.12968/hosp.2002.63.3.2058. PMID 11933816
- [Background] Andrews FJ, Griffiths RD. Glutamine: essential for immune nutrition in the critically ill. Br J Nutr. 2002 Jan;87 Suppl 1:S3-8. doi: 10.1079/bjn2001451. PMID 11895153
- [Background] Griffiths RD. Specialized nutrition support in critically ill patients. Curr Opin Crit Care. 2003 Aug;9(4):249-59. doi: 10.1097/00075198-200308000-00001. PMID 12883278
- [Background] Griffiths RD. Outcome of critically ill patients after supplementation with glutamine. Nutrition. 1997 Jul-Aug;13(7-8):752-4. doi: 10.1016/s0899-9007(97)83039-0. PMID 9263282
- [Background] Griffiths RD, Jones C, Palmer TE. Six-month outcome of critically ill patients given glutamine-supplemented parenteral nutrition. Nutrition. 1997 Apr;13(4):295-302. PMID 9178278
- [Background] Yeh CL, Hsu CS, Yeh SL, Lin MT, Chen WJ. Dietary glutamine supplementation reduces cellular adhesion molecule expression and tissue myeloperoxidase activity in mice with gut-derived sepsis. Nutrition. 2006 Apr;22(4):408-13. doi: 10.1016/j.nut.2005.10.007. Epub 2006 Feb 3. PMID 16458482
- [Background] Singleton KD, Beckey VE, Wischmeyer PE. GLUTAMINE PREVENTS ACTIVATION OF NF-kappaB AND STRESS KINASE PATHWAYS, ATTENUATES INFLAMMATORY CYTOKINE RELEASE, AND PREVENTS ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) FOLLOWING SEPSIS. Shock. 2005 Dec;24(6):583-9. doi: 10.1097/01.shk.0000185795.96964.71. PMID 16317391
- [Background] Wischmeyer PE, Kahana M, Wolfson R, Ren H, Musch MM, Chang EB. Glutamine induces heat shock protein and protects against endotoxin shock in the rat. J Appl Physiol (1985). 2001 Jun;90(6):2403-10. doi: 10.1152/jappl.2001.90.6.2403. PMID 11356807
- [Background] Wischmeyer PS, Serkova KN: Glutamine attenuates multiple pathways of sepsis-induced injury and improves survival following peritonitis: role of heat stress protein pathway manipulation. Presented at Society for Critical Care Medicine 2004.
- [Background] Ziegler TR, Ogden LG, Singleton KD, Luo M, Fernandez-Estivariz C, Griffith DP, Galloway JR, Wischmeyer PE. Parenteral glutamine increases serum heat shock protein 70 in critically ill patients. Intensive Care Med. 2005 Aug;31(8):1079-86. doi: 10.1007/s00134-005-2690-5. Epub 2005 Jun 23. PMID 15973519
- [Background] Singleton KD, Serkova N, Beckey VE, Wischmeyer PE. Glutamine attenuates lung injury and improves survival after sepsis: role of enhanced heat shock protein expression. Crit Care Med. 2005 Jun;33(6):1206-13. doi: 10.1097/01.ccm.0000166357.10996.8a. PMID 15942332
- [Background] Zhou YP, Jiang ZM, Sun YH, Wang XR, Ma EL, Wilmore D. The effect of supplemental enteral glutamine on plasma levels, gut function, and outcome in severe burns: a randomized, double-blind, controlled clinical trial. JPEN J Parenter Enteral Nutr. 2003 Jul-Aug;27(4):241-5. doi: 10.1177/0148607103027004241. PMID 12903886
- [Background] De-Souza DA, Greene LJ. Intestinal permeability and systemic infections in critically ill patients: effect of glutamine. Crit Care Med. 2005 May;33(5):1125-35. doi: 10.1097/01.ccm.0000162680.52397.97. PMID 15891348
- [Background] Garrel D, Patenaude J, Nedelec B, Samson L, Dorais J, Champoux J, D'Elia M, Bernier J. Decreased mortality and infectious morbidity in adult burn patients given enteral glutamine supplements: a prospective, controlled, randomized clinical trial. Crit Care Med. 2003 Oct;31(10):2444-9. doi: 10.1097/01.CCM.0000084848.63691.1E. PMID 14530749
- [Background] Dechelotte P, Hasselmann M, Cynober L, Allaouchiche B, Coeffier M, Hecketsweiler B, Merle V, Mazerolles M, Samba D, Guillou YM, Petit J, Mansoor O, Colas G, Cohendy R, Barnoud D, Czernichow P, Bleichner G. L-alanyl-L-glutamine dipeptide-supplemented total parenteral nutrition reduces infectious complications and glucose intolerance in critically ill patients: the French controlled, randomized, double-blind, multicenter study. Crit Care Med. 2006 Mar;34(3):598-604. doi: 10.1097/01.CCM.0000201004.30750.D1. PMID 16505644
- [Background] Bakalar B, Duska F, Pachl J, Fric M, Otahal M, Pazout J, Andel M. Parenterally administered dipeptide alanyl-glutamine prevents worsening of insulin sensitivity in multiple-trauma patients. Crit Care Med. 2006 Feb;34(2):381-6. doi: 10.1097/01.ccm.0000196829.30741.d4. PMID 16424718
- [Background] Goeters C, Wenn A, Mertes N, Wempe C, Van Aken H, Stehle P, Bone HG. Parenteral L-alanyl-L-glutamine improves 6-month outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2032-7. doi: 10.1097/00003246-200209000-00013. PMID 12352037
- [Background] Wischmeyer PE, Lynch J, Liedel J, Wolfson R, Riehm J, Gottlieb L, Kahana M. Glutamine administration reduces Gram-negative bacteremia in severely burned patients: a prospective, randomized, double-blind trial versus isonitrogenous control. Crit Care Med. 2001 Nov;29(11):2075-80. doi: 10.1097/00003246-200111000-00006. PMID 11700398
- [Background] Mertes N, Schulzki C, Goeters C, Winde G, Benzing S, Kuhn KS, Van Aken H, Stehle P, Furst P. Cost containment through L-alanyl-L-glutamine supplemented total parenteral nutrition after major abdominal surgery: a prospective randomized double-blind controlled study. Clin Nutr. 2000 Dec;19(6):395-401. doi: 10.1054/clnu.2000.0142. PMID 11104589
- [Background] Ockenga J, Borchert K, Rifai K, Manns MP, Bischoff SC. Effect of glutamine-enriched total parenteral nutrition in patients with acute pancreatitis. Clin Nutr. 2002 Oct;21(5):409-16. doi: 10.1054/clnu.2002.0569. PMID 12381339
- [Background] He Xian-li, Ma Qing-jiu, Lu Jian-guo, Chu Yan-kui, Du Xi-lin: Effect of total parenteral nutrition (TPN) with and without glutamine dipeptide supplementation on outcome in severe acute pancreatitis (SAP). Clinical Nutrition supp 2004; 1: 43 - 47.
- [Background] Burnham EL, Moss M, Ziegler TR. Myopathies in critical illness: characterization and nutritional aspects. J Nutr. 2005 Jul;135(7):1818S-1823S. doi: 10.1093/jn/135.7.1818S. PMID 15987872
- [Background] Biolo G, De Cicco M, Dal Mas V, Lorenzon S, Antonione R, Ciocchi B, Barazzoni R, Zanetti M, Dore F, Guarnieri G. Response of muscle protein and glutamine kinetics to branched-chain-enriched amino acids in intensive care patients after radical cancer surgery. Nutrition. 2006 May;22(5):475-82. doi: 10.1016/j.nut.2005.11.003. Epub 2006 Feb 10. PMID 16472976
- [Background] van den Berg A, van Elburg RM, Westerbeek EA, Twisk JW, Fetter WP. Glutamine-enriched enteral nutrition in very-low-birth-weight infants and effects on feeding tolerance and infectious morbidity: a randomized controlled trial. Am J Clin Nutr. 2005 Jun;81(6):1397-404. doi: 10.1093/ajcn/81.6.1397. PMID 15941893
- [Background] Schulman AS, Willcutts KF, Claridge JA, Evans HL, Radigan AE, O'Donnell KB, Camden JR, Chong TW, McElearney ST, Smith RL, Gazoni LM, Farinholt HM, Heuser CC, Lowson SM, Schirmer BD, Young JS, Sawyer RG. Does the addition of glutamine to enteral feeds affect patient mortality? Crit Care Med. 2005 Nov;33(11):2501-6. doi: 10.1097/01.ccm.0000185643.02676.d3. PMID 16276173
- [Background] Neu J, Roig JC, Meetze WH, Veerman M, Carter C, Millsaps M, Bowling D, Dallas MJ, Sleasman J, Knight T, Auestad N. Enteral glutamine supplementation for very low birth weight infants decreases morbidity. J Pediatr. 1997 Nov;131(5):691-9. doi: 10.1016/s0022-3476(97)70095-7. PMID 9403648
- [Background] Poindexter BB, Ehrenkranz RA, Stoll BJ, Wright LL, Poole WK, Oh W, Bauer CR, Papile LA, Tyson JE, Carlo WA, Laptook AR, Narendran V, Stevenson DK, Fanaroff AA, Korones SB, Shankaran S, Finer NN, Lemons JA; National Institute of Child Health and Human Development Neonatal Research Network. Parenteral glutamine supplementation does not reduce the risk of mortality or late-onset sepsis in extremely low birth weight infants. Pediatrics. 2004 May;113(5):1209-15. doi: 10.1542/peds.113.5.1209. PMID 15121931
- [Background] Rao XP, Zhu LQ, Lian HH. [Protective effects of glutamine on the intestinal mucosal barrier in young rabbits under hemorrhagic shock]. Zhongguo Dang Dai Er Ke Za Zhi. 2006 Feb;8(1):66-70. Chinese. PMID 16522245
- [Background] Neu J, Afzal A, Pan H, Gallego E, Li N, Li Calzi S, Caballero S, Spoerri PE, Shaw LC, Grant MB. The dipeptide Arg-Gln inhibits retinal neovascularization in the mouse model of oxygen-induced retinopathy. Invest Ophthalmol Vis Sci. 2006 Jul;47(7):3151-5. doi: 10.1167/iovs.05-1473. PMID 16799062
- [Background] Tian H, Wang KF, Wu TJ. [Effect of total parenteral nutrition with supplementation of glutamine on the plasma diamine oxidase activity and D-lactate content in patients with multiple organ dysfunction syndrome]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2006 Oct;18(10):616-8. Chinese. PMID 17038253
- [Background] Ali S, Roberts PR. Nutrients with immune-modulating effects: what role should they play in the intensive care unit? Curr Opin Anaesthesiol. 2006 Apr;19(2):132-9. doi: 10.1097/01.aco.0000192800.95172.47. PMID 16552219
- [Background] Alpers DH. Glutamine: do the data support the cause for glutamine supplementation in humans? Gastroenterology. 2006 Feb;130(2 Suppl 1):S106-16. doi: 10.1053/j.gastro.2005.11.049. PMID 16473057
- [Background] Jiang H, Chen W, Hu W, Cai B, Liao RJ. [The impact of glutamine-enhanced enteral nutrition on clinical outcome of patients with critical illness: a systematic review of randomized controlled trials]. Zhonghua Shao Shang Za Zhi. 2009 Oct;25(5):325-30. Chinese. PMID 19951553
- [Background] Friedman LM. Fundamentals of clinical trials. 3th ed. New York: Springer;1998.
- [Background] Koletzko B, Goulet O, Hunt J, Krohn K, Shamir R; Parenteral Nutrition Guidelines Working Group; European Society for Clinical Nutrition and Metabolism; European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN); European Society of Paediatric Research (ESPR). 1. Guidelines on Paediatric Parenteral Nutrition of the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) and the European Society for Clinical Nutrition and Metabolism (ESPEN), Supported by the European Society of Paediatric Research (ESPR). J Pediatr Gastroenterol Nutr. 2005 Nov;41 Suppl 2:S1-87. doi: 10.1097/01.mpg.0000181841.07090.f4. No abstract available. PMID 16254497